CLINICAL TRIAL: NCT07259525
Title: Escitalopram Plasma Concentrations in Premenopausal and Postmenopausal Women
Acronym: MENO-ES
Status: Not yet recruiting | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Imran Gokcen Yilmaz-Karaman, Associate professor doctor, Eskisehir Osmangazi University
Other Study IDs: EskisehirOU 09.09.2025/22
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Therapeutic Drug Monitoring (TDM); Menopause; Depression - Major Depressive Disorder; General Anxiety Disorder
Keywords: escitalopram; desmethylescitalopram; menopause; therapeutic drug monitoring; major depressive disorder; general anxiety disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Premenopausal Women: Women aged 40-60 years, premenopausal, diagnosed with major depressive disorder and/or generalized anxiety disorder, and currently receiving escitalopram treatment.
- Postmenopausal Women: Women aged 40-60 years, postmenopausal, diagnosed with major depressive disorder and/or generalized anxiety disorder, and currently receiving escitalopram treatment.

SUMMARY:
This observational cross-sectional case-control study aims to evaluate the effects of menopausal status on escitalopram metabolism in women. The study will include premenopausal and menopausal women aged 40-60 years who are currently receiving escitalopram treatment and have applied to the Psychiatry Clinic of Eskişehir Osmangazi University. The study aims to identify pharmacokinetic differences associated with hormonal status and to investigate their potential clinical implications. Findings from this research are expected to contribute to the development of evidence-based, individualized treatment strategies for women in menopausal transition.

DETAILED DESCRIPTION:
Participants' plasma escitalopram and desmethylescitalopram levels, mental disorder severity, anthropometric measurements, bioimpedance, CYP2C19 genotype analysis, estradiol and follicle-stimulating hormone (FSH) levels, and corrected QT interval (QTc) length will be assessed. In the preliminary analysis, participants carrying the CYP2C19*1 allele will be selected from the data of 78 participants for comparative analyses. Those with the dominant allele will be selected for final analyses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40 years or older and 60 years or younger
* Diagnosed with major depressive disorder and/or generalized anxiety disorder by an independent psychiatrist (not a member of the research team)
* Prescribed escitalopram treatment by an independent psychiatrist (not a member of the research team)
* Receiving escitalopram treatment for at least one month and on a stable dose for at least one week
* Willing to participate in the study and provide informed consent
* Additional inclusion criterion for the menopausal group: Amenorrhea for at least one year (consistent with menopause diagnosis)
* Additional inclusion criteria for the premenopausal group: Having regular menstrual cycles and being in the luteal phase (within 14 days after ovulation) of the menstrual cycle

Exclusion Criteria:

* Diagnosis of intellectual disability, dementia, psychotic disorders, schizoaffective disorder, or bipolar disorder
* Alcohol or substance use disorder
* Diagnosis of hepatic failure, renal failure, or cardiac failure
* Severe malnutrition
* Presence of an active systemic infectious or inflammatory disease
* Current use of hormone replacement therapy for menopause
* Use of oral contraceptives
* Pregnancy or breastfeeding
* Use of medications known to affect escitalopram plasma concentration
* Use of medications that affect the CYP2C19 enzyme
* Detection of alleles other than the predominant CYP2C19*1 genotype in genetic analyses

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Eligibility is restricted to participants assigned female at birth, as the study focuses on premenopausal and menopausal physiological status.
Study Population: Participants are women aged 40 to 60 years who have been diagnosed with major depressive disorder and/or generalized anxiety disorder and are currently receiving escitalopram treatment. All participants were recruited from the Psychiatry Clinic of Eskişehir Osmangazi University.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Dose-Related Plasma Escitalopram Concentrations | Up to 14 days
  Plasma escitalopram concentrations will be measured in participants using therapeutic drug monitoring methods. The primary objective is to compare dose-related plasma escitalopram concentrations between premenopausal and menopausal women receiving escitalopram treatment.
Metabolite to Drug Ratios | Up to 14 days
  Plasma escitalopram and desmethylescitalopram concentrations will be measured in participants using therapeutic drug monitoring methods. The primary objective of the study is to evaluate differences in drug metabolism by comparing metabolite-to-parent drug ratios between premenopausal and menopausal women receiving escitalopram.
Association between plasma S-desmethylescitalopram/escitalopram ratio and serum estradiol levels | Up to 14 days
  The primary outcome is the evaluation of the relationship between the plasma S-desmethylescitalopram/escitalopram metabolite-to-parent drug ratio and serum estradiol concentrations in all participants. The study will test whether lower estradiol levels are associated with higher metabolite-to-drug ratios.

CONTACTS AND LOCATIONS:
Overall Officials: İmran G Yılmaz Karaman, Associtate Professor Doctor, Principal Investigator — Eskişehir Osmangazi University, Faculty of Medicine
Locations (1):
- Eskişehir Osmangazi University, Faculty of Medicine, Department of Psychiatry, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Participants' data will be stored anonymously in an online data repository. IPD will be shared as a study report after data completion is finished.
Supporting Information: CSR
Time Frame: We plan to finish data collection in January 2028, and we plan to publish IPD in 6 months after that.
Access Criteria: IPD will be open to the public.
URL: https://osf.io/